CLINICAL TRIAL: NCT03174574
Title: Two Cancers, One Gene
Brief Title: Two Cancers, One Gene. Why Some People in Families Develop Melanoma or Pancreas Cancer, While Still Others Never Develop Cancer.
Acronym: TCOG
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Gloria M. Petersen, Principal Investigator, Mayo Clinic
Other Study IDs: 16-005414; R01CA208517 (NIH)
Record Dates: First submitted 2017-05-31; First posted 2017-06-02 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Pancreas Cancer; Melanoma
MeSH Terms: conditions — Pancreatic Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Whole blood, serum, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Individuals who are affected with pancreas cancer and melanoma as well as those without either cancer who have been identified as 1st or 2nd degree relatives of family members with pancreas cancer and melanoma will be asked to participate. The participant will be asked to complete a survey about their health and family history of cancer and to give a blood sample for specific gene testing and storage for future research studies.The overall goal of this study is to understand the factors that increase susceptibility and expression of pancreatic cancer and melanoma in high risk families.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are affected with pancreas cancer and melanoma as well as those without either cancer who have been identified as 1st or 2nd degree relatives of family members with pancreas cancer and melanoma.

Exclusion Criteria:

* Under the age of 18, Non-English speaking or unable to provide informed consent, inmates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants and family members of participants currently enrolled under IRB #354-06 and #355-06 who have been identified as members of a family with at least one blood related relative with pancreas cancer, and there is a known mutation carrier of CDKN2A. Some of the family members may have previously enrolled in IRB protocol #354-06 or #355-06; others may not have ever participated in research.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
Genomic and risk factor differences among family members who share identical predisposing CDKN2A gene mutations, with different phenotypes; will discover patterns of tumorigenesis, tissue specificity, gene-gene, and gene-environment interactions. | Each participant provides a research blood sample and completes a questionnaire.This is the duration of their the participant's direct involvement. The duration of generating genotypes and analysis of risk factors may extend up to two years.
  Genotypes of potential modifier genes will be identified in multiple kindreds that feature pancreatic cancer and melanoma and known to carry CDKN2A germline mutations. The investigators will then determine common germline variants in potential CDKN2A mutant carriers using targeted sequencing and search for genetic modifiers by performing Illumina HumanOmni5Exome-4 Beadchip with Infinium LCG on germline DNA. The Illumina microarray contains over 4.5 million markers, of which 528,675 are exonic, and includes over 2.6 million SNPs that would be considered common. The investigators will analyze the genetic and risk factor data collected through the completed surveys by participants using both statistical genetic and machine learning methods. As a means of extension and potential validation, the investigators will then similarly study up to 200 members who are mutation carriers in 39 other CDKN2A mutation-positive kindreds.

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Petersen, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials